CLINICAL TRIAL: NCT07181954
Title: CT-based Radiomics for Prediction of MIT Family Translocation Kidney Cancer: a Multicenter, Retrospective Clinical Study
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA, ECFAH of FMU [2025]794
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: Renal Cell Carcinoma; Computed Tomography; MIT
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project intends to construct a multicenter retrospective study, retrospectively collect clinical, imaging, pathological and prognostic data of patients, establish a complete data management system, establish a prediction model based on CT radiomics characteristics by combining radiomics, and verify the internal and external sequence of the model, which will improve the preoperative clinical diagnosis level of MIT family translocation kidney cancer, and then guide personalized and precise diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of RCC;
2. Have complete clinical, pathological and follow-up data;
3. Renal CT plain scan and enhanced images can be obtained from the image storage and transmission system (PACS)

Exclusion Criteria:

1. Patients who are not suitable for treatment: patients with severe comorbidities or unable to receive any form of treatment;
2. Combined with other malignant tumors: have been treated with other malignant tumors (or have other untreated active malignancies at the same time);
3. Patients with poor CT image quality/absence;
4. Patients with missing clinical/pathological/follow-up data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective data collection was conducted from January 2009 to December 2023 at the First Affiliated Hospital of Fujian Medical University, the Provincial Hospital Affiliated to Fuzhou University, the Second Affiliated Hospital of Fujian Medical University, the First Affiliated Hospital of Chongqing Medical University, and the First Affiliated Hospital of Xiamen University.
Sampling Method: Probability Sample
Enrollment: 746 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative renal tumor pathological diagnosis type | 1 week

IPD SHARING:
Plan to Share IPD: No